CLINICAL TRIAL: NCT04623619
Title: Use of Acetyl L-Carnitine in Patients With Covid-19 Pneumonia
Brief Title: Efficacy and Safety of Acetyl L-Carnitine in COVID-19 Patients With Mild-to-Moderate Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo (Other)
Responsible Party: Principal Investigator, Antonio Cascio, Direttore UOC Malattie Infettive e Tropicali, Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20201109
Record Dates: First submitted 2020-11-09; First posted 2020-11-10 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Covid19
Keywords: acetyl L-Carnitine
MeSH Terms: conditions — COVID-19 | interventions — Acetylcarnitine

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, open-label, controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetyl L-Carnitine (Experimental): Acetyl L-Carnitine
  Interventions: Dietary Supplement: Acetyl L-Carnitine
- Standard of care (No Intervention): Standard of care

INTERVENTIONS:
Dietary Supplement: Acetyl L-Carnitine — Administering 2 gr of Acetyl L-Carnitine orally in addition to the standard of care therapy for 14 days
  Arms: Acetyl L-Carnitine

SUMMARY:
Different studies showed that acetyl L-Carnitine (LC) positively affects the development and maturation of T lymphocytes, involved in the immune response to viral agents. It also contributes to the inhibition of ROS production and to the remodulation of the cytokine network typical of the systemic inflammatory syndrome.

Given the potential protective effects of LC, it is suggested as a supportive and therapeutic option in patients with coronavirus infection. Given this background, in the light of the current COVID-19 emergency, it is the intention of the investigators to conduct a prospective, randomized, open-label, controlled study in the cohort of hospitalized patients with covid-19 pneumonia, administering 2 gr of LC orally in addition to the standard of care therapy (SOC).

The investigators hypothesize that the use of LC will be associated with an earlier improvement of clinical and biohumoral parameters after 14 days of LC treatment when compared to the group of patients provided with standard care.

DETAILED DESCRIPTION:
Different studies showed that acetyl L-Carnitine (LC) positively affects the development and maturation of T lymphocytes, involved in the immune response to viral agents. It also contributes to the inhibition of ROS production and to the remodulation of the cytokine network typical of the systemic inflammatory syndrome.

SARS-CoV-2 virus activates the human cell ACE2 receptor, triggering a series of deleterious events. In COVID19, renin-angiotensin is upregulated and the pathway is overexpressed and a progressive cytokine storm is always observed. In all these pathogenic processes, LC could play a modifier function to enhance condition. LC can be beneficial to the antioxidant effects of Angiotensin II by inhibiting NF-kB and down-regulating NOX1and NOX2. For LC, an anti-apoptotic and genome-stabilizer role was estimated by inhibiting pro-apoptotic caspases and activating PARP-1. LC is an immunomodulator that downregulates pro-inflammatory cytokines including TNF-α, IL-6, and IL-1 that could extinguish the cytokine storm. LC can also serve as a protective agent against COVID19 cardiotoxicity due to disruption in the ACE2-mediated signaling pathway, cytokine storm, pulmonary dysfunction, and side effects of medications.

In patients with coronavirus infection, provided LC's possible protective effects, it is suggested as a supportive and therapeutic alternative.

Given this background, in the light of the current COVID-19 emergency, it is the intention of the investigators to conduct a prospective, randomized, open-label, controlled study in the cohort of hospitalized patients with covid-19 pneumonia, administering 2 gr of LC orally in addition to the standard of care therapy (SOC).

The investigators hypothesize that the use of LC will be associated with an earlier improvement of clinical and humoral parameters after 14 days of LC treatment when compared to the group of patients provided with standard care.

ELIGIBILITY:
Inclusion Criteria:

* Positive swab test of SARS-CoV-2
* Pneumonia related to SARS-CoV-2
* Signature of informed consent

Exclusion Criteria:

* Unsigned informed consent
* Negative swab test of SARS-CoV-2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-15 (Estimated); Primary Completion 2021-04-29 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | 72 hours
  Change of hospital mortality

SECONDARY OUTCOMES:
C reactive protein (CRP) levels | 72 hours
  Reduction of CRP levels > 50% in comparison with CRP levels at the admission, within 72 hours after the administration
IL-6 levels | 72 hours
  Reduction of IL-6 levels > 50% in comparison with IL-6 at the admission, within 72 hours after the administration
D-dimer levels | 72 hours
  Reduction of D-dimer levels > 50% in comparison with D-dimer at the admission, within 72 hours after the administration
Hospital stay | up to 24 weeks
  Length of hospital stay
Duration of positive PCR swab | 5 days
  Time length of negativization of PCR molecular swab

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Cascio, MD, PhD, Principal Investigator — University of Palermo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blanca AJ, Ruiz-Armenta MV, Zambrano S, Miguel-Carrasco JL, Gonzalez-Roncero FM, Fortuno A, Revilla E, Mate A, Vazquez CM. l-Carnitine ameliorates the oxidative stress response to angiotensin II by modulating NADPH oxidase through a reduction in protein kinase c activity and NF-kappaB translocation to the nucleus. Food Chem. 2017 Aug 1;228:356-366. doi: 10.1016/j.foodchem.2017.02.011. Epub 2017 Feb 6. PMID 28317735
- [Background] Puskarich MA, Kline JA, Krabill V, Claremont H, Jones AE. Preliminary safety and efficacy of L-carnitine infusion for the treatment of vasopressor-dependent septic shock: a randomized control trial. JPEN J Parenter Enteral Nutr. 2014 Aug;38(6):736-43. doi: 10.1177/0148607113495414. Epub 2013 Jul 12. PMID 23851424
- [Background] Diao B, Wang C, Tan Y, Chen X, Liu Y, Ning L, Chen L, Li M, Liu Y, Wang G, Yuan Z, Feng Z, Zhang Y, Wu Y, Chen Y. Reduction and Functional Exhaustion of T Cells in Patients With Coronavirus Disease 2019 (COVID-19). Front Immunol. 2020 May 1;11:827. doi: 10.3389/fimmu.2020.00827. eCollection 2020. PMID 32425950
- [Background] Moretti S, Alesse E, Di Marzio L, Zazzeroni F, Ruggeri B, Marcellini S, Famularo G, Steinberg SM, Boschini A, Cifone MG, De Simone C. Effect of L-carnitine on human immunodeficiency virus-1 infection-associated apoptosis: a pilot study. Blood. 1998 May 15;91(10):3817-24. PMID 9573019
- [Background] Wang ZY, Liu YY, Liu GH, Lu HB, Mao CY. l-Carnitine and heart disease. Life Sci. 2018 Feb 1;194:88-97. doi: 10.1016/j.lfs.2017.12.015. Epub 2017 Dec 11. PMID 29241711
- [Background] Mohammadi M, Hajhossein Talasaz A, Alidoosti M. Preventive effect of l-carnitine and its derivatives on endothelial dysfunction and platelet aggregation. Clin Nutr ESPEN. 2016 Oct;15:1-10. doi: 10.1016/j.clnesp.2016.06.009. Epub 2016 Jun 27. PMID 28531771
- [Background] Gorlinger K, Dirkmann D, Gandhi A, Simioni P. COVID-19-Associated Coagulopathy and Inflammatory Response: What Do We Know Already and What Are the Knowledge Gaps? Anesth Analg. 2020 Nov;131(5):1324-1333. doi: 10.1213/ANE.0000000000005147. PMID 33079850